CLINICAL TRIAL: NCT01749371
Title: Vitamin E Supplementation in Burned Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Shriners Hospitals for Children (Other); Memorial Hermann Hospital (Other); University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12-189
Record Dates: First submitted 2012-12-10; First posted 2012-12-13 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Burn
Keywords: Alpha-Tocopherol; Inflammation; Oxidative Stress; Malondialdehyde; Isoprostanes; Lung Dysfunction; Wound Healing
MeSH Terms: conditions — Burns; Inflammation | interventions — Vitamin E; alpha-tocopheryl nicotinate; alpha-Tocopherol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early Vitamin E (Experimental): Vitamin E is administered from Days 1-15 after the initial excision surgery after admission.
  Interventions: Drug: Vitamin E
- Delayed Vitamin E (Experimental): Vitamin E is administered from Days 16-30 after the initial excision surgery after admission.
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: Vitamin E — 1200 IU dl-alpha tocopheryl acetate after the initial excision surgery after admission (days 1-15 or days 16-30)
  Other Names: dl-Alpha Tocopheryl; Alpha Tocopherol; Aqueous Vitamin E Oral Drops

SUMMARY:
A dietary antioxidant, alpha-tocopherol, will be used to potentially attenuate Vitamin E short- and long-term losses in plasma and adipose, reverse the oxidative stress of burn injury and, in the process, decrease the secondary consequences of burn injury, including lung injury and impaired wound healing. This may improve the quality of life of the burn patient by preventing pathophysiology that may result from oxidative stress and may reduce hospital stay. Our research will lay the foundation for the future development of effective, safe, and economic therapeutic interventions to treat burn injury-associated metabolic abnormalities. Also, it will provide the basis for the development of supplemental regulations and pharmacotherapy to treat burn patients with vitamin E. The risks are very reasonable in relation to the anticipated benefits to our subjects because a) vitamin E is a simple vitamin that is abundant and approved for clinical use, and b) the subjects will be monitored consistently for the minimal increased tendency to bleed.

DETAILED DESCRIPTION:
Please see above.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 - 85 years
* ≥40% total body surface area burn

Exclusion Criteria:

* Septic shock
* Bleeding disorders
* Diabetes, or on diabetes medications or anti-lipidemic agents
* Arthritis
* Known kidney/renal disease, endocrine disease, cancer, heart disease, osteoporosis, liver disease
* Congestive heart failure
* Positive hepatitis or HIV screens
* Pregnancy (women)

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Plasma Alpha- and Gamma-Tocopherol | Days 0-30
  Plasma measurements of alpha- and gamma-tocopherol as an indicator of antioxidant status

SECONDARY OUTCOMES:
Pulmonary Function Testing | Day 30
  Assessment of pulmonary function by measuring variables such as functional vital capacity of the lungs and volume ventilation in an effort-dependent exam
Exercise Stress Test | Day 30
  Assessment of strength and cardiopulmonary function through use of exercise
Wound Healing | Days 0-30
  Assessment of variables of the wound such as redness and scar height
Plasma and Urine Malondialdehyde, Isoprostanes, Vitamin E Metabolites | Days 0-30
  Assessment of antioxidant and oxidant status in plasma (short-term)
Adipose Alpha- and Gamma-Tocopherol | Days 0-30
  Assessment of antioxidant and oxidant status in adipose (long-term)

CONTACTS AND LOCATIONS:
Overall Officials: Perenlei Enkhbaatar, MD, PhD, Principal Investigator — University of Texas; Linda E Sousse, PhD, MBA, Study Director — University of Texas
Locations (3):
- United States (3):
  - University of Texas Southwestern Medical Center, Parkland Health and Hospital System, Dallas, Texas
  - University of Texas Medical Branch: Blocker Burn Unit and Shriners Hospitals for Children, Galveston, Texas
  - Memorial Hermann Hospital Burn Intensive Care Unit, Houston, Texas